CLINICAL TRIAL: NCT03597581
Title: A Phase 1 Study of RGX-202-01 (Ompenaclid) , a Small Molecule Inhibitor of the Creatine Transporter SLC6a8, as a Single Agent and as Combination Therapy in Patients With Advanced Gastrointestinal Malignancies With Select Expansion Cohorts
Brief Title: A Study of RGX-202-01 (Ompenaclid) as Combination Therapy in RAS Mutant Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inspirna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGX-202-001
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Cancer; Gastrointestinal Neoplasms; Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma; Gastric Cancer; Gastric Neoplasm; KRAS Mutation-Related Tumors; CRC; Colorectal Cancer Metastatic
Keywords: SLC6a8; Creatine transporter; FOLFIRI; Colorectal Cancer; CRC; KRAS; Colorectal Cancer Metastatic; NRAS; RAS; FOLFOX
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms | interventions — IFL protocol; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single agent Ompenaclid (RGX-202-01) Dose Escalation (Experimental): Ompenaclid (RGX-202-01) is administered orally twice or three times daily on days 1-28 of each 28-day cycle. The dose regimen is dependent on the cohort in which the patient is enrolled.
  Interventions: Drug: ompenaclid
- Ompenaclid (RGX-202-01) in combination with FOLFIRI Dose Escalation (Experimental): Ompenaclid (RGX-202-01) is administered orally twice or three times daily on days 1-28 of each 28-day cycle. The dose regimen is dependent on the cohort in which the patient is enrolled.
  FOLFIRI is administered as follows: irinotecan 180 mg/m2 intravenously over 90 minutes concurrently with folinic acid (leucovorin) 400 mg/m2 intravenously over 2 hours, followed by 5-FU 400 mg/m2 intravenous bolus and then 5-FU 2400 mg/m2 intravenous infusion over 46 hours, on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: ompenaclid; Drug: FOLFIRI
- Expansion: 2nd Line Colorectal Cancer (CRC) KRAS (+) (Experimental): 2nd Line CRC RAS (+)
  Ompenaclid (RGX-202-01) is administered orally twice on days 1-28 of each 28-day cycle.
  FOLFIRI is administered as follows: irinotecan 180 mg/m2 intravenously over 90 minutes concurrently with folinic acid (leucovorin) 400 mg/m2 intravenously over 2 hours, followed by 5-FU 400 mg/m2 intravenous bolus and then 5-FU 2400 mg/m2 intravenous infusion over 46 hours, on Days 1 and 15 of each 28-day cycle.
  Bevacizumab is administered as follows: 5 mg/kg on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: ompenaclid; Drug: FOLFIRI; Drug: Bevacizumab
- Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Escalation (Experimental): RGX-201-01 is administered orally twice or three times daily on days 1-28 of each 28-day cycle. The dose regimen is dependent on the cohort in which the patient is enrolled.
  The FOLFOX regimen used for this protocol consists of oxaliplatin given at 85 mg/m2 IV together with leucovorin at 400 mg/m2 IV (substitution with levo-leucovorin 200 mg/m2 IV is allowed) (duration per institutional policy), followed by a 5-FU bolus of 400 mg/m2 (over 2-5 minutes), and then continuous infusional 5-FU given at a dose of 2400 mg/m2 over 46-48 hours (1200 mg/m2/day), given on Days 1 and 15 of each 28-day cycle. A minimum of 8 FOLFOX cycles should be received if tolerated per standard of care guidelines.
  Interventions: Drug: ompenaclid; Drug: Bevacizumab; Drug: FOLFOX regimen
- Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Expansion (Experimental): Ompenaclid (RGX-202-01) is administered orally twice or three times daily on days 1-28 of each 28-day cycle. The dose regimen is dependent on the cohort in which the patient is enrolled.
  The FOLFOX regimen used for this protocol consists of oxaliplatin given at 85 mg/m2 IV together with leucovorin at 400 mg/m2 IV (substitution with levo-leucovorin 200 mg/m2 IV is allowed) (duration per institutional policy), followed by a 5-FU bolus of 400 mg/m2 (over 2-5 minutes), and then continuous infusional 5-FU given at a dose of 2400 mg/m2 over 46-48 hours (1200 mg/m2/day), given on Days 1 and 15 of each 28-day cycle. A minimum of 8 FOLFOX cycles should be received if tolerated per standard of care guidelines.
  Interventions: Drug: ompenaclid; Drug: Bevacizumab; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: ompenaclid — RGX-202-01 (ompenaclid) is a small molecule inhibitor of the creatine transporter, SLC6a8.
  Other Names: RGX-202-01
Drug: FOLFIRI — FOLFIRI is a chemotherapy regimen consisting of irinotecan, leucovorin, and 5-fluorouracil. Irinotecan is a topoisomerase inhibitor, which prevents DNA from uncoiling and duplicating.
  Arms: Expansion: 2nd Line Colorectal Cancer (CRC) KRAS (+); Ompenaclid (RGX-202-01) in combination with FOLFIRI Dose Escalation
Drug: Bevacizumab — Bevacizumab is a vascular endothelial growth factor inhibitor.
  Arms: Expansion: 2nd Line Colorectal Cancer (CRC) KRAS (+); Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Escalation; Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Expansion
Drug: FOLFOX regimen — The FOLFOX regimen used for this protocol consists of oxaliplatin given at 85 mg/m2 IV together with leucovorin at 400 mg/m2 IV (substitution with levo-leucovorin 200 mg/m2 IV is allowed) (duration per institutional policy), followed by a 5-FU bolus of 400 mg/m2 (over 2-5 minutes), and then continuous infusional 5-FU given at a dose of 2400 mg/m2 over 46-48 hours (1200 mg/m2/day), given on Days 1 and 15 of each 28-day cycle. A minimum of 8 FOLFOX cycles should be received if tolerated per standard of care guidelines
  Arms: Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Escalation; Ompenaclid (RGX-202-01) in combination with FOLFOX Dose Expansion

SUMMARY:
This is a Phase 1 study currently evaluating PO administered ompenaclid in combination with FOLFIRI and bevacizumab in patients with advanced (i.e., locally advanced and unresectable, or metastatic) previously treated colorectal adenocarcinoma. The single agent ompenaclid dose escalation stage and the ompenaclid in combination with FOLFIRI and bevacizumab dose escalation stage of the study has been completed; the expansion stage of ompenaclid in combination with FOLFIRI and bevacizumab is ongoing. In April-24 a protocol amendment added a new dose escalation and expansion stage which will evaluate ompenaclid in combination with FOLFOX and bevacizumab in patients with metastatic CRC. It is anticipated that a total of 30 patients will be enrolled in this new dose escalation and expansion stage of the study.

DETAILED DESCRIPTION:
Expansion Stage: Ompenaclid in Combination with FOLFIRI and Bevacizumab

Eligible patients must have had PD after receiving only one prior regimen considered standard of care for CRC in the advanced/metastatic setting, which must have been an oxaliplatin-containing regimen. However, if the patient has mismatch repair deficient (dMMR)/ microsatellite instability-high (MSI-H) CRC, they must have also received prior treatment with pembrolizumab or a US Food and Drug Administration (FDA) approved PD-1/PD-L1 inhibitor. Patients who developed recurrent metastatic CRC within 12 months of completion of adjuvant oxaliplatin and 5-FU based therapy are also eligible as long as they did not receive an additional first-line regimen in the advanced/metastatic setting.

All patients will receive ompenaclid at a dose of 2400 mg or 3000 mg administered PO BID on a continuous daily schedule. The FOLFIRI dose and schedule will be irinotecan 180 mg/m2 IV over 90 minutes concurrently with leucovorin 400 mg/m2 IV over 2 hours, followed by 5-FU 2400 mg/m2 IV infusion over 46 hours, on Days 1 and 15 of each 28-day cycle, and the bevacizumab dose will be 5 mg/kg on Days 1 and 15 of each 28-day cycle.

The goal of the expansion stage will be to provide further characterization of the efficacy, safety and tolerability of combination therapy, and PK and pharmacodynamics of ompenaclid when combined with FOLFIRI and bevacizumab, at two different dose levels of ompenaclid. The dose of ompenaclid in combination with FOLFIRI and bevacizumab in the expansion stage will be 2400 or 3000 mg PO BID. The 3000 mg BID dose represents the last dose of ompenaclid that has been evaluated in combination with FOLFIRI and bevacizumab in the dose escalation stage and which was not considered to be the MTD. Approximately 52 patients will be treated with ompenaclid in combination with FOLFIRI and bevacizumab, all of whom had/will have CRC.

Dose Escalation and Expansion Stages: Ompenaclid in Combination with FOLFOX and Bevacizumab

Based on experience from the completed single agent and combination therapy dose escalation parts of this study where an MTD was not reached and no DLTs were observed, the dose escalation of ompenaclid in combination with FOLFOX and bevacizumab will evaluate 3 escalating doses of ompenaclid (1800 mg [Cohort 1], 2400 mg [Cohort 2], and 3000 mg [Cohort 3] administered BID PO) on Days 1-28 of a 28-day cycle, in combination with FOLFOX and bevacizumab dosing.

Dose escalation will follow a standard 3+3 design. All safety data from all patients enrolled in each cohort will be reviewed by a Safety Review Committee (SRC) to confirm any DLTs that were experienced and to make a determination regarding enrollment in the next cohort. A patient must have received at least 70% of their total planned ompenaclid doses and both the courses of FOLFOX and bevacizumab planned during the 28-day DLT assessment period with follow-up through the end of this period to be eligible for DLT assessment. If a DLT necessitates enrollment of additional patients into a cohort, all of the safety data for that cohort will be reviewed by the SRC after those additional patients have completed the DLT assessment period.

The goal of the expansion stage will be to provide further characterization of safety and tolerability of combination therapy, and PK and pharmacodynamics of ompenaclid when combined with FOLFOX and bevacizumab at two different dose levels of ompenaclid: the MTD/maximum tested dose as determined in the dose escalation stage, and one dose level below the MTD/maximum tested dose.

A total of approximately 30 patients will be treated with ompenaclid in combination with FOLFOX plus bevacizumab to provide characterization of the safety and tolerability of combination therapy, and PK and pharmacodynamics of ompenaclid when combined with FOLFOX plus bevacizumab. This total includes approximately 10 patients treated at each of the two ompenaclid dose levels during the expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have histologic or cytologic evidence of a RAS colorectal cancer of adenocarcinoma or poorly differentiated histology and must have disease that is resistant to or relapsed following available standard systemic therapy or for which there is no standard systemic therapy or reasonable therapy likely to result in clinical benefit or if such therapy has been refused by the patient.
* The patient must have advanced disease, defined as cancer that is either metastatic or locally advanced and unresectable (and for which additional radiation therapy or other locoregional therapies are not considered feasible).
* Pathologically documented adenocarcinoma or poorly differentiated locally advanced/metastatic colorectal cancer
* Have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the Investigator
* Adults ≥18 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 1
* Adequate cardiac function, as defined by left ventricular ejection fraction (LVEF) ≥45%
* Adequate organ function
* Prothrombin time ≤1.5 x ULN or international normalized ratio within ≤1.5; and either partial thromboplastin time or activated partial thromboplastin time ≤1.5 x ULN. Patients on warfarin may be included if on a stable dose with a therapeutic INR <3.5

Inclusion Criteria for RGX-202-01 plus FOLFIRI and bevacizumab expansion stages:

For the expansion stage only, patients must have a tumor that is laboratory-confirmed to be RAS mutant.

* Must have received only one prior standard of care oxaliplatin-containing regimen for locally advanced/metastatic colorectal cancer (CRC)
* Must have received prior treatment with pembrolizumab or an FDA approved PD-1/L1 inhibitor as well, if the patient has dMMR/MSI-H colorectal cancer
* May have received prior treatment with bevacizumab, cetuximab, or panitumumab, or an FDA approved biosimilar.

Exclusion Criteria for RGX-202-01 plus FOLFIRI and bevacizumab expansion stages:

* Unresolved Grade > 2 toxicities from prior anticancer therapy; excluding Grade 2 chemotherapy-related neuropathy, alopecia; and excluding Grade 2-3 asymptomatic laboratory abnormalities if considered clinically insignificant by the Investigator, or can be managed with available medical therapies
* Has malignancy of small cell, neuroendocrine, or squamous histology
* Unable to meet the requirement of an adequate treatment washout period before enrollment
* Has additional malignancy that may confound the assessment of study endpoints. Participants with non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, and melanoma in situ), organ-confined prostate cancer with no evidence of progressive disease are not excluded
* Has clinically significant cardiovascular disease (New York Heart Association Class III or IV congestive heart failure, history of myocardial infarction, uncontrolled angina, unstable angina or stroke within 6 months before enrollment, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication
* Has clinically active brain or leptomeningeal metastases
* Has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding
* Has an ongoing chronic hepatopathy of any origin
* Has an evidence of muscular dystrophies or ongoing muscle pathology
* Has oxygen-support requirements
* Has corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (males)
* Has a physical abnormality or medical condition that limits swallowing multiple pills or has a history of non-adherence to oral therapies
* Has a malabsorption condition, such as short bowel syndrome, impaired GI function or GI disease that may significantly alter absorption, or a high likelihood of impending bowel obstruction, such as strictures
* Has clinically significant ascites (i.e. requiring paracentesis within the preceding 28 days or treatment with pain medication)
* Has a medical condition which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities

Exclusion Criteria for RGX-202-01 plus FOLFIRI and bevacizumab dose escalation and expansion stages:

* Has known dihydropyrimidine dehydrogenase (DPD) deficiency or is on treatment with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine, within 4 weeks prior to the start of treatment
* Has known homozygous or heterozygous for UGT1A1*28, UGT1A1*6, UGT1A9*1 or ABCG2 allele
* Require treatment with strong CYP3A4 inhibitors or strong UGT1A1 inhibitors
* Previously treated with FOLFIRI or other irinotecan containing regimens
* Has proteinuria ≥ 2gm/24 and/or nephrotic syndrome. Patients with a proteinuria 2+ or greater urine dipstick reading should undergo further assessment, e.g., a 24-hour urine collection
* History of acute or subacute intestinal occlusion - except if such an event occurred only around the time of diagnosis - or chronic inflammatory bowel disease or chronic diarrhea
* History of severe, non-healing wounds, ulcers or bone fractures
* History of arterial thromboemboli or severe hemorrhage within 6 months of prior FOLFIRI treatment with an exception of tumor bleeding before tumor resection surgery
* History of hemorrhagic diathesis or tendency towards thrombosis

Inclusion Criteria: FOLFOX/Bevacizumab Combination

To be enrolled in this substudy, patients must meet all of the following criteria during the screening period:

1. The patient has signed informed consent prior to initiation of any study-specific procedures or treatment.
2. The patient must have previously untreated metastatic colorectal adenocarcinoma, defined as cancer that is metastatic and for which additional radiation therapy or other locoregional therapies in curative intent are not considered feasible or beneficial. Note that patients who have had previous systemic anticancer therapy as neoadjuvant or adjuvant therapy and had a metastatic recurrence at least 12 months after the last dose of adjuvant oxaliplatin will also be eligible.
3. The patient must have a tumor that is laboratory-confirmed to be RAS-mutant based on the tumor tissue analysis. RAS-mutant status confirmation by liquid biopsy is acceptable only if the tumor sample is not available. For patients with newly diagnosed disease, RAS-mutant status must be obtained before initiation of therapy.
4. The patient must have disease that is measurable by standard imaging techniques by RECIST version 1.1 or by physical examination methods (ruler or calipers). For patients with prior radiation therapy, measurable lesions must be outside of any prior radiation field(s), unless disease progression has been documented at that disease site subsequent to radiation.
5. The patient is ≥ 18 years old.
6. The patient has an ECOG Performance Score of ≤ 1.
7. The patient has adequate baseline organ function, as demonstrated by the following:

   1. Serum creatinine ≤ 1.5 x institutional ULN and calculated creatinine clearance > 50 mL/minute;
   2. Serum albumin ≥ 2.5 g/dl;
   3. Bilirubin ≤ 1.5 x institutional ULN or ≤ 2.5 x institutional ULN for patients with known Gilbert's disease;
   4. AST and ALT ≤ 2.5 x institutional ULN; patients with hepatic metastases may have AST and ALT ≤ 5 x institutional ULN;
   5. ANC ≥ 2.0 x 109/L;
   6. Hemoglobin ≥ 8 g/dL and no RBC transfusions during 14 days before the start of study treatments;
   7. Platelet count ≥ 100 x 109/L and no platelet transfusions during 14 days before the start of study treatments.
8. For patients not taking anticoagulation therapy: INR ≤ 1.5 or PT ≤ 1.5 x ULN; and either PTT or aPTT ≤ 1.5 x ULN. Patients on warfarin/anticoagulation therapy may be included if on a stable dose with a therapeutic anticoagulation range.
9. The patient has a LVEF ≥ 45% as determined by either ECHO or MUGA scanning.
10. If the patient is a WOCBP, she has had a negative serum or urine pregnancy test within 2 weeks prior to treatment.
11. Men and WOCBP agree to use acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for at least 6 months after the last dose of bevacizumab or 2 months after the last dose of ompenaclid, whichever is later.
12. The patient is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria: FOLFOX/Bevacizumab Combination

Potential patients to be enrolled in the FOLFOX/bevacizumab combination phase of this study who meet any of the following criteria during the screening period will be excluded:

1. Patients who have received neoadjuvant or adjuvant FOLFOX chemotherapy and have development of metastatic disease documented within 12 months after completion of oxaliplatin.

   • Patients may have received prior single agent fluoropyrimidine therapy if administered for the purpose of radiosensitization or as a single systemic agent (if the development of metastatic disease is documented at least 12 months from completion of neoadjuvant/adjuvant therapy).
2. Any Grade neurotoxicity.
3. Patients who have dMMR/MSI-H CRC.
4. The patient has received treatment with chemotherapy, biological therapy, external-beam radiation, or other systemic anticancer therapy within 12 months prior to the administration of study treatments (42 days for prior nitrosourea or mitomycin-C).
5. Known allergy or hypersensitivity to platinum-containing medications, 5-FU or leucovorin.
6. Has an additional active malignancy that may confound the assessment of the study endpoints. Patients with a past cancer history with substantial potential for recurrence must be discussed with the Medical Monitor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, and melanoma in situ), organ-confined prostate cancer with no evidence of PD (Gleason ≤ 6).
7. Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure (see Section 13), uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension (defined as SBP > 160 mmHg or DBP > 90 mmHg), or clinically significant arrhythmias not controlled by medication).
8. History of arterial thromboembolism or severe hemorrhage within 6 months prior to inclusion in the study, with the exception of tumor bleeding before tumor resection surgery.
9. Known or suspected active brain or leptomeningeal metastases. Pre-existing asymptomatic brain or leptomeningeal metastases should be stable with no need for steroid therapy. If the patient has had prior radiation, the washout for metastases or brain surgery is 14 days before the start of treatment. CNS imaging is not required prior to study entry unless there is a clinical suspicion of CNS involvement.
10. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant or breast -eeding.
12. Ongoing chronic hepatopathy of any origin.
13. Clinically significant ascites (i.e., requiring paracentesis within the prior 28 days or medical treatment for abdominal pain).
14. Evidence of muscular dystrophies or ongoing muscle pathology.
15. Oxygen-support requirements.
16. QTcF > 450 msec (males) or > 470 msec (females).
17. Physical abnormality or medical condition that limits swallowing multiple pills or has a history of non-adherence to oral therapies.
18. Gastrointestinal disorder(s) that would significantly impede the absorption of an oral agent.
19. Known DPD deficiency or is on treatment with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine, within 4 weeks prior to the start of treatment.
20. Marked proteinuria (≥ 2 g/24 h) and/or nephrotic syndrome. Patients with a proteinuria 2 + or greater on urinalysis/urine dipstick reading should undergo further assessment, e.g., a 24-hour urine collection.
21. Severe, non-healing wounds, ulcers or bone fractures.
22. History of hemorrhagic diathesis or tendency towards thrombosis that is not optimally managed.
23. Medical condition not listed above which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
RGX-202-01 maximum tolerated dose | 6 months
  Maximum tolerated dose (MTD), or the maximum tested dose at which multiple dose-limiting toxicities (DLTs) are not observed, of RGX-202-01 as a single agent, and separately, in combination with FOLFIRI +/- bevacizumab.
RGX-202-01 overall response rate | 24 months
  Overall response rate (ORR) associated with RGX-202-01 treatment in combination with FOLFIRI plus bevacizumab.
RGX-202-01 treatment-emergent adverse events | 24 months
  Number of participants with treatment-emergent adverse events (TEAEs) with severity as determined by CTCAE v5 associated with RGX-202-01 treatment as a single agent, and separately, in combination with FOLFIRI +/- bevacizumab.

SECONDARY OUTCOMES:
RGX-202-01 maximum plasma concentration | 24 months
  Pharmacokinetics: Maximum plasma concentration (Cmax) of RGX-202-01.
RGX-202-01 area under the curve | 24 months
  Pharmacokinetics: Area under the curve (AUC) of RGX-202-01.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wasserman, MD, Study Chair — CMO
Locations (17):
- United States (17):
  - Arizona Oncology Associates, PC - HAL, Prescott Valley, Arizona
  - Arizona Oncology Associates, PC - HOP E, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sharp HealthCare, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - UCLA Department of Medicine, Santa Monica, California
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, P.A, McAllen, Texas
  - Texas Oncology, P.A, Tyler, Texas